CLINICAL TRIAL: NCT06576297
Title: Novel Respiratory Training as Part of Palliative Care for Older Adults With Heart Failure
Acronym: RETRO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: The Pittsburgh Foundation (Other)
Responsible Party: Principal Investigator, Daniel Forman, MD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY23010048
Record Dates: First submitted 2024-02-22; First posted 2024-08-28 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Aging; Heart Failure With Preserved Ejection Fraction; Heart Failure With Reduced Ejection Fraction; Frailty; Physical Function; Quality of Life
Keywords: 70 and older; Inspiratory Muscle Training; Heart Failure with Preserved Ejection Fraction; Heart Failure with Reduced Ejection Fraction; Frailty; Physical function; Quality of life
MeSH Terms: conditions — Frailty | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator, Outcomes assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Participants in the usual care group will be telephoned at 4 and 8 weeks, and AE/SAE will be reviewed.
  Interventions: Other: Standard of Care
- IMT Group: Inspiratory Muscle Training (IMT) (Experimental): IMT exercise sessions addition to standard of care.
  Interventions: Other: Inspiratory Muscle Training (IMT)

INTERVENTIONS:
Other: Inspiratory Muscle Training (IMT) — IMT using a PrO2™ inspiratory training device will incorporate the Test of Incremental Respiratory Endurance (TIRE)9 technology to achieve an optimized exercise training regimen.
  Arms: IMT Group: Inspiratory Muscle Training (IMT)
Other: Standard of Care — Standard of Care Participants in the usual care group will be telephoned at 4 and 8 weeks, and AE/SAE will be reviewed.
  Arms: Standard of Care

SUMMARY:
In a randomized controlled trial, to study the utility of inspiratory muscle training (IMT) to improve functional outcomes in adults aged ≥70 years with heart failure (HF) who have been referred to palliative care for end-stage HF management.

* The study team hypothesize that older HF patients will be able to use IMT safely, reliably, and effectively in a 12-week home-based training regimen.
* The study team hypothesize that physical function (sit to stand, gait speed, grip strength), respiratory/pulmonary function, self-efficacy, fatigue and quality of life will increase among older HF patients randomized IMT versus those randomized to usual care.

DETAILED DESCRIPTION:
Heart failure (both HF with reduced ejection fraction [HFrEF] and HF with preserved ejection fraction [HFpEF]) are on the rise in our aging population. Exercise intolerance is a leading detriment of the disease. While it is understood that exercise training is beneficial, strategies to achieve exercise training in this population are inherently limited, particularly as the issues that contribute to HF pathophysiology (i.e., advanced age, frailty, multimorbidity) also predispose to sedentariness, weakening, frailty, sarcopenia, fatigue, and cognitive impairment. Physical activity and particularly exercise training may be hard to initiate and sustain especially because it is encumbered by limitations. Home-based exercise training strategies are conceptually appealing in respect to practicality of access, but the associated issues of monitoring for effective and safe exercise, motivation, and tracking of training are all difficult to achieve in a home-based format. Furthermore, many older adults lack suitable space or resources for traditional home-based exercise training.

IMT with the PrO2™ device responds to these challenges with a novel approach to achieve physiologically robust training effect (strength training of the diaphragm) in a way that mitigates breathlessness and augments multiple indices of function in a way that is practical and safe, even at home. The electronic dimensions of the device also enable embedded trackability and behavioral prompts. Overall, this is a novel approach to a common, familiar problem, and it responds directly to a well-known problem of dyspnea, sedentariness and related functional decline that undermines current standards of HF care.

Existing models of exercise training for HF rely primarily on site-based regimens of aerobic and strength training modalities. Implementation barriers include unfeasible logistics for patients who often do not drive, particularly as many older patients struggle with frailty as well as limitations due to cognitive decline, sensory impairment, and/or socioeconomic challenges amidst the predictable complexities associated with advanced age. Fear and poor motivation compound these limitations, with limited options to motivate, supervise, and track progress for many candidates.

This proposal promotes the concept of "Palliative Care Rehab" which is transformational in concept. It shifts the premise of cardiac rehabilitation from cardiorespiratory fitness to more rudimentary goals of activities of daily living and self-efficacy. Likewise, rather than focusing on traditional cardiovascular endpoints of exercise testing and high performance, this study is oriented to submaximal endpoints, fatigability, and qualitative metrics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Advanced Heart Failure (HFrEF or HFpEF), with NYHA class II, III, or IV despite a minimum of
* 6 weeks of treatment
* Age >70 years
* Male and Female
* Optimal therapy according to AHA/ACC and HFSA HF guidelines

Exclusion Criteria:

* Patients living in an institutional setting (e.g., skilled nursing home) during the intended period of this study.
* Major cardiovascular event or procedure within the prior 6 weeks.
* HF secondary to significant uncorrected primary valvular disease (except mitral regurgitation secondary to left ventricular dysfunction). If valve replacement has been performed, the participant may not be enrolled for 12 months after this procedure.
* Dementia
* Severe COPD (FEV1<50%), PVD, and/or Anemia
* End-stage malignancy
* Severe valvular heart disease
* Psychiatric hospitalization within the last 3 months
* Chronic ETOH or drug dependency.

We will exclude all of the following special populations:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Safety of a 12-week home-based IMT program. | Baseline and weekly for 12 weeks
  AE/SAE (IMT vs. controls): number Completion of the 3-month intervention (IMT vs. controls)

SECONDARY OUTCOMES:
Adherence to IMT training sessions | Baseline and weekly for 12 weeks
  Number of IMT sessions competed over 12-week intervention
Improvement in MIP | Baseline, 12 weeks
  Improvement in MIP (IMT vs. controls): cm H2O
Sit to stand | Baseline, 12 weeks
  5-times Sit-to-Stand: seconds
Gait speed | Baseline, 12 weeks
  4 m Gait Speed: m/sec
Grip strength | Baseline, 12 weeks
  Grip Strength: pounds
Self-efficacy | Baseline, 12 weeks
  Self-efficacy: Sullivan Self-Efficacy; 0-52; higher score is more favorable
Quality of Life | Baseline, 12 weeks
  Quality of Life: Kansas City Cardiomyopathy Questionnaire (KCCQ): score 0-100; higher is more favorable than lower score.
Fatigue | Baseline, 12 weeks
  Fatigue: PROMIS Item Bank v1.0 - Fatigue - short form 13a (FACIT-Fatigue): scale 0-52; lower indicates less fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E. Forman, M.D, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Hope to publish results of this pilot study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available one year after study is closed.
Access Criteria: Per PI discretion